CLINICAL TRIAL: NCT06226402
Title: Comparative Study Between the Effect of Nebulized and Intravenous Hypertonic Saline 3% on the Management of Patients With Acute Respiratory Distress Syndrome
Brief Title: Effect of Nebulized and Intravenous Hypertonic Saline 3% on the Management of Patients With Acute Respiratory Distress Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Elsayed Mohamed Elfakhrany, Resident of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36264MS225/6/23
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Nebulization; Hypertonic Saline; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Saline Solution, Hypertonic; Nebulizers and Vaporizers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): Patients will receive the standard pharmacotherapy of Acute Respiratory Distress Syndrome (ARDS) patients.
- Inhalational group (Experimental): Patients will receive the standard pharmacotherapy + hypertonic saline 3% (5ml) nebulizer /8hr.
  Interventions: Drug: Hypertonic saline 3% nebulizer
- Intravenous group (Experimental): Patients will receive the standard pharmacotherapy + hypertonic saline 3% intravenous over 24 hours to maintain plasma Na level between 145-150 mEq/L.
  Interventions: Drug: Intravenous hypertonic saline 3%

INTERVENTIONS:
Drug: Hypertonic saline 3% nebulizer — Patients will receive the standard pharmacotherapy + hypertonic saline 3% (5ml) nebulizer /8hr.
  Arms: Inhalational group
Drug: Intravenous hypertonic saline 3% — Patients will receive the standard pharmacotherapy + hypertonic saline 3% intravenous over 24 hours to maintain plasma Na level between 145-150 mEq/L.
  Arms: Intravenous group

SUMMARY:
The aim of our study is to compare between the effect of nebulized and intravenous injection of hypertonic saline 3% on the outcome of patients with acute respiratory distress syndrome.

DETAILED DESCRIPTION:
Acute Respiratory Distress Syndrome (ARDS) is a life threatening form of respiratory failure, characterized by acute, diffuse, inflammatory lung injury that results in increased alveolar capillary permeability and the development of non-hydrostatic pulmonary edema.

Clinically, ARDS manifests as marked hypoxemia and respiratory distress; patients often progress to respiratory failure that requires invasive mechanical ventilation in the intensive care unit.

No specific pharmacological treatment is available for ARDS, which is associated with high morbidity and mortality. The mainstay of therapy in ARDS is supportive therapy and invasive mechanical ventilation based on lung-protective strategies using low tidal volume (VT) at 4-6 ml/kg of predicted body weight (PBW) and plateau pressure (p PLAT) below 30 cm H2O, but other adjunctive therapies have been trialed with various degrees of efficacy, including neuromuscular blockade, prone positioning, recruitment maneuvers (RMs), vasodilators, and extracorporeal membrane oxygenation (ECMO).

Hypertonic saline 3% NaCl with 513 mEq/L of Na and 513 mEq/L of Cl is a potent anti-inflammatory agent, and immunomodulator, which exerts inhibitory effects in several stages of the inflammatory cascade. Hypertonic saline, at a cellular level, decreases alveolar macrophage activation, polymorph nuclear leucocyte recruitment, priming and activation, as well as cell surface adhesion molecule expression. High plasma sodium contributes to high plasma osmolality which can be lung protective and would seem to be a logical choice for treatment of ARDS.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 to 60 years old.
* Both sexes.
* Patients with mild and moderate ARDS whose PaO2/FiO2 ratio ≥ 150 according to the Berlin definition of Acute Respiratory Distress Syndrome.

Exclusion Criteria:

* Refusal to participate in the study.
* Malignancy.
* Patients on chemotherapy.
* Decompensated renal, hepatic and cardiac disease.
* Patients with hypernatremia whose serum Na above 155 mEq/L.
* Patients with ARDS whose PaO2/FiO2 ratio > 150.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who will need mechanical ventilation | 28 days after intervention
  Number of patients who will need mechanical ventilation will be assessed.

SECONDARY OUTCOMES:
Length of ICU stay | 28 days after intervention
  Length of ICU stay will be measured from the admission till the discharge from the hospital.
Lung injury score (Murray score) | 24 hours after intervention
  Murray score (lung injury score) will be calculated daily in the morning based on information obtained from:
  1. Number of quadrants of infiltrations from chest X-ray.
  2. Hypoxic index.
  3. Positive end expiratory pressure (PEEP) required on the ventilator to get better oxygenation.
  4. Static compliance.
Incidence of mortality | 28 days after intervention
  Incidence of mortality will be assessed at 7th, and 28th day.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.